CLINICAL TRIAL: NCT02900261
Title: Comparison of Methods to Measure the Consumption of Sodium and Caffeine in Children
Brief Title: Study on Sodium and Caffeine in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Hôpital du Valais (Other); Federal Food Safety and Veterinary Office (Unknown)
Responsible Party: Principal Investigator, Arnaud Chiolero, Epidemiologist & Senior lecturer, University of Lausanne Hospitals
Other Study IDs: 2016-01178
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Sodium; Caffeine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — This study is observational and does not entail any intervention. Different methods to assess sodium and caffeine consumption will be compared.

SUMMARY:
This study will compare different methods (24 hour urine collection, evening and morning spots, and questionnaires) to measure the consumption of sodium and cafeine in children and adolescents.

DETAILED DESCRIPTION:
Sodium consumption among adults is high in Switzerland, as in most parts of the world. It is expected to be high in children as well, but little is still known. 24 hour urine collection is the golden standard to assess sodium consumption. However, this method is logistically difficult, especially for children. Therefore, alternatives are needed. Urinary spots have been used as a proxy to estimate sodium excretion over 24 hour in adults, but not in children. This study will assess whether urinary spots can be used to estimate sodium consumption in children in comparison to 24 hour urine collections.

Caffeine consumption has risen in children over the past years, mainly before of the increase in consumption of soda drinks. A precise way to measure caffeine consumption is by assessing the concentration of caffeine and its metabolites in 24 hour urine samples. An alternative to 24 hour urine collection is using questionnaires, however this remains difficult due to the multiples food sources of caffeine. This study will compare caffeine consumption estimated by 24 hour urine collection and by a semi-quantitative food frequency questionnaire targeting caffeine containing products.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 and 16 years of age

Exclusion Criteria:

* A sickness that affects the consumption and excretion of sodium and caffeine (for example, diabetes, cardiovascular or gastrointestinal problems, chronic kidney disease, renal insufficiency)
* Taking medication that affects sodium excretion (for example, diuretics)
* A intravenous perfusion during the urine collection
* Insufficient knowledge of French to understand the instructions

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 6 and 16 years of age, following ambulatorily at the Hospital of Sion
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Urinary sodium excretion | Over a 2-day period
  Measured in 24 hour urine and estimated from 3 different urinary spots
Urinary caffeine and related metabolites excretion | Over a 2-day period
  Measured in 24 hour urine and estimated by a semi-quantitative food frequency questionnaire

SECONDARY OUTCOMES:
Sodium consumption | Over a 2-day period
  Estimated by a semi-quantitative food frequency questionnaire
Urinary phosphate excretion | Over a 2-day period
  Measured in 24 hour urine and estimated from 3 different urinary spots
Urinary caffeine and metabolites excretion | Over a 2-day period
  Measured in 24 hour urine and estimated from 3 different urinary spots
Urinary albumine excretion | Over a 2-day period
  Measured in 24 hour urine and estimated from 3 different urinary spots
Urinary protein excretion | Over a 2-day period
  Measured in 24 hour urine and estimated from 3 different urinary spots

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Chiolero, MD PhD, Principal Investigator — arnaud.chiolero@chuv.ch
Locations (1):
- Hôpital du Valais, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be published in an article. The full dataset will be made available in the DATA@IUMSP repository, http://data.iumsp.ch.

REFERENCES:
- [Derived] Paccaud Y, Rios-Leyvraz M, Bochud M, Tabin R, Genin B, Russo M, Rossier MF, Bovet P, Chiolero A, Parvex P. Spot urine samples to estimate 24-hour urinary calcium excretion in school-age children. Eur J Pediatr. 2020 Nov;179(11):1673-1681. doi: 10.1007/s00431-020-03662-z. Epub 2020 May 9. PMID 32388721
- [Derived] Rios-Leyvraz M, Bochud M, Tabin R, Genin B, Russo M, Rossier MF, Eap CB, Bovet P, Chiolero A. Monitoring caffeine intake in children with a questionnaire and urine collection: a cross-sectional study in a convenience sample in Switzerland. Eur J Nutr. 2020 Dec;59(8):3537-3543. doi: 10.1007/s00394-020-02187-3. Epub 2020 Feb 3. PMID 32016643
- [Derived] Rios-Leyvraz M, Bovet P, Tabin R, Genin B, Russo M, Rossier MF, Bochud M, Chiolero A. Urine Spot Samples Can Be Used to Estimate 24-Hour Urinary Sodium Excretion in Children. J Nutr. 2018 Dec 1;148(12):1946-1953. doi: 10.1093/jn/nxy211. PMID 30517722
- [Derived] Rios-Leyvraz M, Bovet P, Bochud M, Genin B, Russo M, Rossier MF, Tabin R, Chiolero A. Estimation of salt intake and excretion in children in one region of Switzerland: a cross-sectional study. Eur J Nutr. 2019 Oct;58(7):2921-2928. doi: 10.1007/s00394-018-1845-4. Epub 2018 Oct 19. PMID 30341681